CLINICAL TRIAL: NCT06937021
Title: The Impact of an Art and Philosophy-based Intervention on Children's Eco-anxiety: A Pilot Study
Brief Title: The Impact of an Art and Philosophy-based Intervention on Children's Eco-anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bishop's University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Catherine Malboeuf-Hurtubise, Associate professor, psychologist, Bishop's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102683
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Eco-anxiety; Psychological Distress; Tolerance to Distress; Hope; Mental Health
Keywords: Art-based interventions; Philosophical inquiry; eco-anxiety; children; schools; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art-based intervention (ABI) (Active Comparator)
  Interventions: Other: Art based intervention (ABI)
- Arts and philosophy intervention (APBI) (Experimental)
  Interventions: Other: Art and philosophy intervention (APBI)

INTERVENTIONS:
Other: Art and philosophy intervention (APBI) — 8 session intervention delivered during school time. Each session involves an art activity with a corresponding philosophical discussion.
  Arms: Arts and philosophy intervention (APBI)
Other: Art based intervention (ABI) — A 8 session intervention delivered during school time. Each session involve a creative arts activity.
  Arms: Art-based intervention (ABI)

SUMMARY:
Objective: To examine the impact of climate change on children's mental health by comparing the effectiveness of an arts only intervention (ABI) and an arts and philosophy-based intervention (APBI) on children's eco-anxiety, tolerance to distress and hope for the future in school settings. The investigators hypothesized that the children assigned to the combined arts and philosophy intervention would show reductions in self-reported eco-anxiety, as well as increases in tolerance to distress and hope for the future in the context of climate change, when compared to children assigned to the arts-only intervention.

Setting: This study is conducted in public primary schools from England. Participants: Participants are students in grades 3 to 6. Main Outcomes and Measures: The primary outcome is self-reported eco-anxiety scores. Secondary outcomes are self-reported tolerance to distress, hope for the future and mental health (depression and anxiety symptoms).

ELIGIBILITY:
Inclusion Criteria:

* being an elementary school student

Exclusion Criteria:

* not being an elementary school student

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eco-anxiety | From enrollment to the end of treatment at 8 weeks
  Self-reported child eco-anxiety
  Hogg Eco-Anxiety Scale Minimum score: 0 Maximum score: 33 Higher scores mean worse outcomes

SECONDARY OUTCOMES:
Tolerance to distress | From enrollment to the end of treatment at 8 weeks
  Self-reported child tolerance to distress
  Distress Intolerance Index for Youth Minimum score: 0 Maximum score: 36 Higher scores mean worse outcomes
Hope | From enrollment to the end of treatment at 8 weeks
  Self-reported child hope
  1 item house scale: Thinking about climate change, how hopeful would you say you are that things will get better in the future? Minimum score: 0 Maximum score: 4 Higher score means a better outcome
Mental health | From enrollment to the end of treatment at 8 weeks
  Self-reported anxiety and depression symptoms
  Selected items from the anxiety and depression subscales of the Behavior Assessment System for Children-III Minimum score: 0
  Maximum score anxiety: 9 Maximum score depression: 15 Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Malboeuf-Hurtubise, PhD, Principal Investigator — Bishop's University
Locations (1):
- Reach2 Academy, NorthStar Academy, Henhurst Ridge, Burton-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No